CLINICAL TRIAL: NCT02033512
Title: NANOSTRUCTURED TRANSDERMAL HORMONE REPLACEMENT THERAPY RELIEVING MENOPAUSAL SYMPTOMS: A CONFOCAL RAMAN SPECTROSCOPY STUDY
Brief Title: TRANSDERMAL HRT RELIEVING POSTMENOPAUSAL SYMPTOMS
Acronym: THRT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Potiguar (Other)
Collaborators: Universidade Federal de Sergipe (Other)
Responsible Party: Principal Investigator, MARCO BOTELHO, PhD, University Potiguar
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNPQ202316; CNPq (Other Grant/Funding Number: CNPq202316/2001-4)
Record Dates: First submitted 2013-12-10; First posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Menopause
Keywords: Post-menopause; Hormone Replacement Therapy; Nanotechnology; Biolipid B2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Transdermal Hormone Replacement Therapy — The Blood samples were collected from the subjects early in the morning after an overnight fast. After serum testing, the identification hormone deficiencies, was determined and then, if necessary, additional transdermal progesterone was prescribed. The patients were evaluated 3 months after THRT treatment protocol.
  All the patients were instructed about how to use the progesterone pump for transdermal application, performed in the presence of an experienced physician, in order to guarantee standardization and correct use of the THRT. Compliance was defined as completing seventy percent or more of the transdermal applications.
  Other Names: Biolipideo/B2®
Drug: Transdermal Nanoformulation — The Blood samples were collected from the subjects early in the morning after an overnight fast. After serum testing, the identification hormone deficiencies, was determined and then, if necessary, additional transdermal hormones were prescribed.
  Other Names: Biolipid/B2, Biolipideo/B2, Evidence Soluções Farmaêuticas
Drug: Transdermal formulation — 66 patients completed the study. In the present analysis, the subjects received daily in the right and left forearm a transdermal nanostructured formulation of Estriol (0.1%) + Estradiol (0.25%) and Progesterone (10%) respectively (Biolipid B2®, Evidence, SP, Brazil) for sixty months. The effects of transdermal hormone formulation were analyzed.
  Other Names: Biolipid/B2®

SUMMARY:
There is a dilemma and a permanent debate about side effects on drugs administered orally. The first-pass metabolism is related with many side effects, since the metabolites of these compounds affect the course of human physiology. Conventional hormone therapy by oral route has been used for relieving menopausal symptoms. Transdermal estrogens have not been used extensively in Brazilian women with menopausal symptomatology, however; recently a previous long term study has indicated no increased risk breast cancer or vasomotor disorders in menopausal women, using transdermal HRT.

DETAILED DESCRIPTION:
This was a prospective long-term clinical trial study of female patients aged 51-70 years old treated for menopause related hormone imbalances. Other results of this study are published elsewhere. Volunteers were recruited from referenced Gynecological Medical service where patient charts are maintained.

This study is a prospective long-term clinical trial study randomized trial assessing the effects of Transdermal HRT on climacteric symptoms and hormone serum levels in early postmenopausal women. Preliminary results of this trial, including the first 42 women enrolled, have been published (3).

In the present analysis, 66 women received daily in the right and left forearms a transdermal nanostructured formulation of Estriol (0.1%) + Estradiol (0.25%) and Progesterone (10%) respectively (Biolipid B2®, Evidence, SP, Brazil) for sixty months. The following were compared: effects of transdermal gel on baseline and after THRT were also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* 1) last menstrual period between 6 months and 3 years before the beginning of the study plus follicle-stimulating hormone (FSH) levels higher than 35 IU/L; 2) age between 51 and 70 years; 3) no use of any medication known to interfere with hormonal levels in the past 6 months.

Exclusion Criteria:

* Patients presenting diabetes, previous hysterectomy, endometrial thickness higher than 5 mm, history of cancer, thromboembolism or established cardio vascular disease were excluded.

Ages: 51 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2003-01; Primary Completion 2004-01 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Estradiol Levels | 5 years
  Effect of Progesterone (10%) associated with Estriol (0.1) +Estradiol (0.25%) Nanoparticles formulation on Estradiol serum levels
  The serum levels of estradiol, over the 60 months of THRT are shown in Figure 8. Statistical analysis of mean Estradiol pretreatment values at baseline was 28.88 ± 39.62 (pg/mL) and after 60 months of THRT showed a significant increase to 51.85 ± 77.50. The data reached a statistical difference (p<0.05) after the treatment with the transdermal formulation.

SECONDARY OUTCOMES:
Effect of Progesterone (10%) associated with Estriol (0.1) +Estradiol (0.25%) Nanoparticles formulation on postmenopausal complaints | 5 years
  The postmenopausal symptomatology analysis of the volunteers subjected to THRT that received the nanoformulation revealed a significant decreasing of postmenopausal scores complaints (Figure 3). These values were statistically significant (P < 0.05), when the mean values from baseline were compared after 60 months of treatment. The extent of satisfaction with the hormone therapy was ~75%. The continuation induced further increases in the extent of satisfaction: 85.2 after one year and 92.5 ± 4.2% at the end of study (P < 0.05).

CONTACTS AND LOCATIONS:
Overall Officials: MARCO A BOTELHO, PhD, Principal Investigator — University Potiguar; Dinalva B Queiroz, MsC, Study Chair — School of Health
Locations (1):
- Gynelogical Center, Fortaleza, Ceará, Brazil

REFERENCES:
- [Derived] Botelho MA, Queiroz DB, Barros G, Guerreiro S, Fechine P, Umbelino S, Lyra A, Borges B, Freitas A, Queiroz DC, Ruela R, Almeida JG, Quintans L Jr. Nanostructured transdermal hormone replacement therapy for relieving menopausal symptoms: a confocal Raman spectroscopy study. Clinics (Sao Paulo). 2014 Feb;69(2):75-82. doi: 10.6061/clinics/2014(02)01. PMID 24519196
- See also: paper published by the research group — http://www.latamjpharm.org/resumenes/31/3/LAJOP_31_3_1_14.pdf